CLINICAL TRIAL: NCT02705599
Title: Stroke Mechanism Evolution in Intracranial Atherosclerotic Stenosis
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Xin Lou, Deputy Chief, Chinese PLA General Hospital
Other Study IDs: HRMRI-NM-Tiantan
Record Dates: First submitted 2016-03-07; First posted 2016-03-10 (Estimated); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Stroke
Keywords: Ischemic stroke; High resolution MRI; Perfusion; Mechanism
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Predictors of the risk of recurrent stroke for patients with symptomatic intracranial atherosclerotic stenosis (ICAS) remain unknown. The study will be to explore the stroke mechanism evolution in patients with ICAS by multi-model magnetic resonance imaging (MRI) which consists of diffusion-weighted imaging (DWI) and high-resolution MRI (HRMRI). The patients with symptomatic ICAS will undergo multi-model MRI. The baseline data, infarct patterns on DWI, and plaque features on HRMRI will be collected. The stroke mechanisms will be determined by the infarct patterns. During the 2 years follow-up, the recurrent ischemic events will be recorded. By comparing the baseline data, infarct patterns, and plaque features in patients with and without recurrent strokes, the high-risk features of patients with symptomatic ICAS will be identified. The evaluation of stroke mechanisms of patients with symptomatic ICAS will be summarized.

DETAILED DESCRIPTION:
Objective:

Primary objective: to identify which plaque features on HRMRI in patients with symptomatic ICAS are related to recurrent stroke.

Secondary objectives: To compare plaque features in subgroups.

Patients enrollment please see Eligibility part.

Methods:

A 3T GE (DISCOVERY MR 750, GE Healthcare, Waukesha, WI, USA) and a 3T Siemens Trio MR scanner (Siemens Healthcare, Ehrlangen, Germany) will be used in this study. The multiple sequences will include 3D time of flight (TOF) MR angiography, 3D T1-weighted imaging, proton attenuation weighted imaging, magnetization-prepared rapid acquisition with gradient-echo sequence (MPRAGE), and contrast enhancement on T1-weighted imaging.

The parameters of multiple sequences on GE MR Scanner are followed. 3D TOF: repetition time (TR) = minimum, echo time (TE) = minimum; field of view (FOV) = 240×220 mm2, matrix = 288×192, slice thickness = 2 mm, flip angle (FA) = 20, and scan time = 1:53 minutes. 3D CUBE T1: TR = 600 ms, TE = minimum, FOV = 240×220 mm2, matrix = 480×480, slice thickness = 0.8 mm, FA = NA, and scan time = 3:33 minutes. 3D CUBE PD: TR = 1500 ms, TE = 40 ms, FOV = 240×220 mm2, matrix = 384×384, slice thickness = 0.8 mm, FA = NA, and scan time = 2:40 minutes. MP RAGE: TR = minimum, TE = 3.3 ms, FOV = 240×240 mm2, matrix = 256×256, slice thickness = 0.8 mm, FA = 12, and scan time = 2:18 minutes.

The parameters of multiple sequences on Siemens MR Scanner are followed. 3D TOF: TR= 24 ms, TE = 4.32 ms; FOV = 140×140 mm2, matrix = 256×256, slice thickness = 0.9 mm, FA = 18, and scan time = 2 min 14 s. 3D SPACE T1: TR = 800 ms, TE = 22 ms, FOV = 180×168 mm2, matrix = 256×251, slice thickness = 0.8 mm, FA = NA, and scan time = 4:4 minutes. 3D SPACE PD: TR = 1700 ms, TE = 23 ms, FOV = 180×180 mm2, matrix = 320×304, slice thickness = 0.6 mm, FA = NA, and scan time = 4:25 minutes. MP RAGE: TR = 776.13 ms, TE = 5.8 ms, FOV = 144×144 mm2, matrix = 240×240, slice thickness = 1 mm, FA = 15, and scan time = 2:39 minutes.

IMAGING EVALUATION In this study, plaques will be identified as focal or diffuse but eccentric wall thickenings compared with normal vessel wall.

Plaque composition will include hemorrhage and calcification. The anatomical location of plaque will be recorded as either one of the four quadrants of the vessel wall on cross-sectional images.

Plaque that is distributed across ≥3 quadrants of the lumen perimeter will be defined as diffuse and that involving ≤2 will be defined as focal.

In this study, enhancement analysis will include both grades and patterns. Enhancement will be classified into 3 different grades: non-enhancement, mild-moderate enhancement, and strong enhancement. Mild-moderate enhancement is defined as less than that of the pituitary infundibulum. Strong enhancement is equal to or stronger than that of the pituitary infundibulum. The pattern of enhancement will be categorized as focal, heterogeneous, or homogenous.

The vessel and wall areas at the maximal lumen narrowing (MLN) site will be measured. The plaque volume will be calculated as the product of the plaque area and the thickness of the slices containing the plaque. The plaque/wall ratio was defined as the plaque area divided by wall area ×100%. The remodeling index was calculated as the ratio of the vessel area at the MLN site to that at the reference site. The reference site was selected based on the Warfarin-Aspirin Symptomatic Intracranial Disease trial method.

STROKE MECHANISMS The stroke includes hypoperfusion, perforator (branch atheromatous disease), artery-to-artery embolism, or co-existing (combinations of these ischemic mechanisms).

FOLLOW-UP At the 2 years follow-up, patients were contacted monthly by phone to determine whether any events had occurred at the first year and three months at the second year. Every three months, patients were examined face-to-face by two neurologists at the first year and every six months at the second year. The follow-up information included transient ischemic attack and ischemic stroke (in any vascular territory), brain hemorrhage, and all-cause death. If these events but death suspected, patients underwent brain computed tomography or MR imaging.

ELIGIBILITY:
Patients suspected of having symptomatic ICAD at admission will be enrolled. All patients will receive a thorough evaluation to determine the cause of their ischemic event (TIA or ischemic stroke), including carotid duplex, transcranial Doppler, echocardiography, electrocardiogram, computed tomography (CT), CT angiography, MRI, magnetic resonance angiography (MRA), or digital subtraction angiography DSA.

Patients will be enrolled in this study according to if they met the following:

* ischemic stroke or TIA in the target territories of the intracranial anterior or posterior circulation within 90 days;
* Lack of coexistent≥50% ipsilateral extracranial carotid artery or vertebral artery stenosis;
* No potential sources of cardio-aortic embolism based on the modified Trial of ORG 10172 in Acute Stroke Treatment classification;
* Age ≥18 years;
* One or more atherosclerotic risk factors including hypertension, hypercholesterolemia, diabetes mellitus, cigarette smoking, and obesity.

Exclusion Criteria:

* Non-atherosclerosis vasculopathy such as vasculitis and arterial dissection diagnosed by comprehensive laboratory work (such as erythrocyte sedimentation rate or C-reactive protein elevations, antinuclear antibody, or antiphospholipid antibody positivity), vascular imaging, and clinical evaluation;
* Contraindication to MR examination, medical instability precluding MR examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Symtomatic patients with intracranial atherosclerostic stenosis
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Ischemic stroke event (in the stenotic vascular territory) | To 2 years
  The primary outcome will include ischemic stroke (in the stenotic vascular territory) and vascular death.

SECONDARY OUTCOMES:
Ischemic stroke event (in the non-stenotic vascular territory) | To 2 years
  The second outcome will include ischemic stroke (in the non-stenotic vascular territory) , transient ischemic attack, brain hemorrhage, and all-cause death.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Lou, M.D. Ph.D., Principal Investigator — Chinese PLA General Hospital; Ning Ma, M.D. Ph.D., Principal Investigator — Beijing Tiantan Hospital
Locations (2):
- China (2):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lyu J, Ma N, Liebeskind DS, Wang DJ, Ma L, Xu Y, Wang T, Miao Z, Lou X. Arterial Spin Labeling Magnetic Resonance Imaging Estimation of Antegrade and Collateral Flow in Unilateral Middle Cerebral Artery Stenosis. Stroke. 2016 Feb;47(2):428-33. doi: 10.1161/STROKEAHA.115.011057. Epub 2016 Jan 5. PMID 26732570
- [Background] Ma N, Jiang WJ, Lou X, Ma L, Du B, Cai JF, Zhao TQ. Arterial remodeling of advanced basilar atherosclerosis: a 3-tesla MRI study. Neurology. 2010 Jul 20;75(3):253-8. doi: 10.1212/WNL.0b013e3181e8e714. PMID 20644151
- [Background] Lopez-Cancio E, Matheus MG, Romano JG, Liebeskind DS, Prabhakaran S, Turan TN, Cotsonis GA, Lynn MJ, Rumboldt Z, Chimowitz MI. Infarct patterns, collaterals and likely causative mechanisms of stroke in symptomatic intracranial atherosclerosis. Cerebrovasc Dis. 2014;37(6):417-22. doi: 10.1159/000362922. Epub 2014 Jul 4. PMID 25011483
- [Derived] Hou Z, Li M, Lyu J, Xu Z, Liu Y, He J, Jing J, Wang R, Wang Y, Lou X, Miao Z, Ma N. Intraplaque Enhancement Is Associated With Artery-to-Artery Embolism in Symptomatic Vertebrobasilar Atherosclerotic Diseases. Front Neurol. 2021 Sep 1;12:680827. doi: 10.3389/fneur.2021.680827. eCollection 2021. PMID 34539546
- [Derived] Yang M, Ma N, Liu L, Wang A, Jing J, Hou Z, Liu Y, Lou X, Miao Z, Wang Y. Intracranial collaterals and arterial wall features in severe symptomatic vertebrobasilar stenosis. Neurol Res. 2020 Aug;42(8):649-656. doi: 10.1080/01616412.2020.1782081. Epub 2020 Jun 23. PMID 32573371
- [Derived] Xu Z, Li M, Lyu J, Hou Z, He J, Mo D, Gao F, Liu X, Sui B, Shen M, Pan Y, Wang Y, Lou X, Miao Z, Luo B, Ma N. Different risk factors in identical features of intracranial atherosclerosis plaques in the posterior and anterior circulation in high-resolution MRI. Ther Adv Neurol Disord. 2020 Mar 13;13:1756286420909991. doi: 10.1177/1756286420909991. eCollection 2020. PMID 32206091
- [Derived] Xu Z, Li M, Hou Z, Lyu J, Zhang N, Lou X, Miao Z, Ma N. Association between basilar artery configuration and Vessel Wall features: a prospective high-resolution magnetic resonance imaging study. BMC Med Imaging. 2019 Dec 26;19(1):99. doi: 10.1186/s12880-019-0388-3. PMID 31878890
- [Derived] Ma N, Xu Z, Lyu J, Li M, Hou Z, Liu Y, Yang M, Mo D, Gao F, Song L, Sun X, Liu L, Liu X, Sui B, Shen M, Ma L, Wang Y, Wang Y, Miao Z, Lou X. Association of Perforator Stroke After Basilar Artery Stenting With Negative Remodeling. Stroke. 2019 Mar;50(3):745-749. doi: 10.1161/STROKEAHA.118.023838. PMID 30661491